# 長庚醫療財團法人林口長庚紀念醫院 受試者同意書



一、計畫名稱:比較 bp-MRI 與 mp-MRI 在 MRI 融合標靶活檢前篩查臨床重要攝護腺癌的隨機對照 試驗

二、研究基本資料

病歷號碼:\_\_\_\_\_

1.計畫編號:

IRB 案號/申請編號: 2311220052

2.試驗(研究)機構:長庚醫療財團法人林口長庚紀念醫院

執行者所屬單位:泌尿腫瘤科

3.委託單位/廠商:長庚醫療財團法人林口長庚紀念醫院

4. 總主持人:馮思中 服務單位:泌尿腫瘤科

職稱:主治醫師 電話:0975365572 共同主持人:王俐人 服務單位:影像診療科

職稱:主治醫師 電話:0975365759

共同主持人:邵翊紘 服務單位:泌尿腫瘤科

職稱:主治醫師 電話:0975361311

協同主持人:莊正鏗 服務單位:泌尿腫瘤科 職稱:主治醫師 電話:0975365573

協同主持人: 虞凱傑 服務單位: 泌尿腫瘤科

職稱:主治醫師 電話:0975366241

協同主持人:林柏宏 服務單位:泌尿腫瘤科

職稱:主治醫師 電話:0975366240

協同主持人:甘弘成 服務單位:泌尿腫瘤科

職稱:主治醫師 電話:0975361365

協同主持人:吳俊德 服務單位:泌尿腫瘤科

職稱:主治醫師 電話:0975360671

協同主持人:黃亮鋼 服務單位:泌尿腫瘤科

職稱:主治醫師 電話:0978835552

受試者 24 小時緊急連絡人與電話: 馮思中醫師 電話: 0975365572 & 03-3281200#7820

5.受試者姓名: 受試者研究編號:

性別: 出生日期:

通訊地址: 聯絡雷話:

## 三、簡介

你好,我們敬邀您參加一個於本院進行之早期攝護腺癌篩檢,對於在雙參數與多參數磁共振成像組中臨床顯著攝護腺癌的檢測情況。依衛生主管機關規定,您必須被告知接受試驗之目的、檢驗及可能的風險。在您同意參加本研究之前,馮思中醫師或其他泌尿科醫師會向您說明這份受試者同意書的內容、回答您的任何疑問,並給予您充分時間考慮,請您再次徹底閱讀這份受試者同意書入職事的問清楚任何問題。此外,要不要參加試驗,完全是自願性質,如果不同意參加試驗,並不會影響到您的正當權益。

四、試驗目的

長庚醫療財團法



本研究的目的是探討在台灣男性中,攝護腺特異性抗原(PSA)水平在 4-20 ng/ml 範圍內且懷疑患 有攝護腺癌時,使用雙參數磁共振成像(bpMRI)與多參數磁共振成像(mpMRI)在檢測和指導針 對臨床顯著攝護腺癌(csPCA)的標靶活檢方面的效果和準確性。此研究旨在比較這兩種 MRI 技術 在確定攝護腺癌標靶活檢位置方面的有效性,以及評估它們對於提高 csPCA 診斷的貢獻程度。通過 這項研究,我們期望能夠為臨床上判斷針對懷疑 csPCA 進行的最佳成像策略提供更明確的指導,從 而提升攝護腺癌診斷和治療的整體效果。

- (1. 雙參數磁共振成像 (bp-MRI) -這是一種用來看身體內部情況的特別照相技術,主要看兩種特殊 圖片來幫助判斷身體是否有病。它能夠快速且較便宜地提供需要的資訊。
- 2. 多參數磁共振成像 (mp-MRI) -這種技術比雙參數磁共振成像來得更詳細,它結合了好幾種不同 的照相方式,為醫生提供更全面的身體內部圖像。這在判斷攝護腺是否有癌症時特別有用。
- 3. 臨床上顯著的攝護腺癌 (csPCA)-指的是那種需要積極治療的攝護腺癌,因為它可能會對健康造 成嚴重影響。)
- 五、納入/排除條件
- 一、如果您符合下列的納入/排除條件才有資格參與本試驗
- 1.納入標準
  - 1. 年龄≥50 歲的男性
  - 2. 臨床上懷疑有攝護腺癌且需進行攝護腺活組織檢查 biopsy
  - 3. 血清攝護腺特異抗原(PSA)水平在 4~20 ng/mL 之間
  - 4. 適合進行磁共振成像(MRI)檢查
  - 5. 直腸指檢 Digital rectal examination, DRE 結果 < cT2 (局限於器官內的癌症)
  - 6. 能夠提供書面知情同意。

(直腸指檢 (DRE)-這是一種醫生用手指檢查肛門和直腸是否有異常的簡單檢查。這項檢查可以幫助 發現攝護腺問題。)

## 2.排除條件

- 1. 在篩檢前 6 個月內有攝護腺活檢(biopsy)史
- 2. 此前已被診斷出攝護腺癌
- 3. 對攝護腺活檢有禁忌症:活動性尿道感染、無法將經直腸超聲探頭插入直腸(腹會陰切 除術、肛門狹窄)、無法矯正的凝血功能障礙、無法停用的抗血小板或抗凝藥物(繼續使 用低劑量阿司匹林在活檢前後是允許的)
- 4. 對磁共振成像檢查有禁忌症:對造影劑過敏、幽閉恐懼症或其他禁忌症(如:腹內金屬
- 5. 由於患者拒絕活檢或在活檢前失訪而沒有攝護腺活檢的組織學結果的患者
- 6. 接受過攝護腺癌治療或任何形式的荷爾蒙治療、免疫治療、化療、盆腔輻射治療的患者
- 7. 撤回本研究知情同意的患者
- 3. 退出標準:
  - 1. 患者無法完成預定的 MRI 檢查
  - 2. MRI 影像品質不足,無法定位臨床顯著攝護腺癌(csPCA)或排除 csPCA 的存在

六、試驗方法與程序說明

目前臨床常規活檢程序,主要依賴經直腸超音波引導的切片檢查,但這一方法在精準度

人體試驗倫理委



頁2之9 版本日期

改進的空間。因此,如何能夠早期且精準地診斷出具有臨床意義的攝護腺癌,成為了一項重要的課題。近期的研究表明,通過結合磁振造影和超音波影像的融合切片檢查技術,可以顯著減少不必要的攝護腺切片檢查,對低風險攝護腺癌的診斷率降低,從而減少了不必要的手術及其可能的併發症。目前,多參數磁振造影(mpMRI)是常用的診斷方法,而本研究將探索一種簡化的雙參數磁振造影(bp-MRI)方法,並將其與傳統的 mpMRI 方法進行比較。

我們計畫預計實施 2 年,受試者來源為臨床科醫師在門診時,懷疑您可能有攝護腺癌且需進一步進行攝護腺活組織檢查時,即可通知主持人或研究相關人員與患者說明,若您若同意參加,需請您簽署同意書。您完成同意書簽署後將依計畫的隨機分派表分派進行 bp-MRI 或 mp-MR,以取得磁振造影參數,攝護腺 MRI 可使用 3.0 特斯拉掃描儀配合盆腔相控陣列線圈進行雙參數和多參數 MRI 攝護腺檢查,無論是否使用對比劑。MRI 結果將根據 PI-RADS (攝護腺成像-報告和數據系統) v2.1 建議報告。MRI 將由有經驗的放射科醫師報告。PI-RADS 3-5 分數將被視為可疑,並將進行針對性加系統性活檢。

# (攝護腺成像報告和數據系統 (PI-RADS)-這是一套幫助醫生用一致的方式解讀攝護腺磁共振成像的規則,讓不同的醫生看圖片時能有相同的理解,幫助提高診斷攝護腺癌的準確性。)

對於在 MRI 上發現可疑病變的患者(在 bp-MRI 或 mp-MRI 上識別為 PI-RADS 3-5 分數的病變), 將通過經會陰部途徑在全麻下進行活檢,每個病變取 3 個針對性活檢核心,另外分別從左右葉取 3 個系統性活檢核心。對於在 MRI 上未識別到可疑病變的患者,將通過經直腸途徑在局部麻醉下進行 標準的 12 核心系統性活檢。所有活檢將由經驗豐富的泌尿科醫師進行,針對性活檢將通過軟件輔 助的 MRI-USG 融合註冊進行。根據我們的臨床指南給予周圍活檢抗生素。

## (MRI-USG 融合技術-這是一種先進的技術,結合了磁共振成像和超聲波掃描,讓醫生能夠更準確地 看到並判斷需要進一步檢查或治療的區域,尤其是在攝護腺癌診斷中。)

患者在攝護腺活檢後如能無重度血尿自行排尿且臨床穩定,則出院。您將在活檢後 10 天內回門診隨訪,審查病理結果和併發症。所有活檢將由經驗豐富的泌尿生殖病理學家評估,並根據國際泌尿病理學會(ISUP)的共識報告。研究期結束於首次回門診隨訪。另外,此 bp-MRI 或 mp-MRI 磁振造影施行地點於本院兒童大樓 B2 磁振造影中心,時間約需要 40-50 分鐘(包含 MRI 前置作業 10-15 分鐘),由取得合格證照之醫放師執行,可做為臨床診斷之用。

## 1.被選為參與者的原因。

- (1) 泌尿科門診之攝護腺癌病人
- (2) 血清攝護腺特異抗原(PSA)水平在 4~20 ng/mL 之間
- (3) 臨床上懷疑有攝護腺癌且需進行攝護腺活組織檢查 biopsy
- (4) **直腸指檢** Digital rectal examination, DRE 結果≤ cT2
- (5) 適合進行磁共振成像(MRI)檢查
- 2.其他依各研究計畫之需要,病歷檢閱、追蹤檢查檢驗或病情資訊相關之重要事項。

## 七、可預期之風險、副作用、發生率及處理方法:

## 1.生理方面:

一般而言,MRI 磁共振成像在身體方面的風險相對較低。它使用磁場和無線電波來創建身體組織的詳細圖像,不涉及離子輻射,通常被認為較安全。然而,存在一些潛在風險或考慮因素,物對別強磁場可能對含鐵或金屬物體造成的影響、使用含鉬對比劑可能引起的過敏反應或其他副作用11·3級. 24 窄空間可能引起的幽閉恐懼症、掃描過程中的噪音不適,以及對於有嚴重腎功能問題的患者最應期間



頁 3 之 9 版本日期

含鉬對比劑可能增加腎性全身性纖維化的風險。

2.心理方面(包含檢體提供者、親屬、族群等):

在本研究中,活檢 biopsy 檢測結果將由您的主治醫師提供詳細解釋。您可能對報告的含義不太明白,或可能因此產生一些與研究計畫無直接關聯的額外疑問。我們會盡力釋解您對檢測結果的任何疑慮,以減少您的擔憂。

3.社會方面(包含檢體提供者、親屬、族群等):

本研究相關人員將盡力保護您提供之資料,您的資料會以編碼標示,並且在未經您同意的情況下,我們不會洩漏任何可能辨認您或您的家人訊息。研究期間所收集的家族史、病歷史、臨床檢驗、實驗數據會分別機密歸檔保存,除非經由您的書面授權或人體試驗委員會同意,否則非研究團隊相關人員無法取得您的個人資料和相關病歷;您的來信詢問也會經由電話跟您做確認後再行答覆。

八、本試驗之禁忌與限制,請您務必要充分配合之事項:

無

九、預期試驗效果

雖然在參與研究期間,您個人可能無法立即受益,但隨著醫藥科技的發展,對於您與您的家人以及 其他社會大眾的健康將會有所助益。

十、緊急狀況之處理

若您參與本研究發生不適之緊急狀況,請隨時與您的主治醫師聯絡,主持人泌尿腫瘤科馮思中醫 師。

試驗主持人24小時聯絡人:馮思中

試驗主持人24小時連絡電話:0975365572。

十一、抽取的檢體將如何處理及儲存地點

無

十二、使用檢體及檢體相關資訊之可能人員

無

十三、預期衍生之商業運用

無

十四、補助、費用負擔與損害補償:

1.補助:無

2. 費用負擔:參加本試驗您不需負擔任何費用

3.損害補償:

- (1)如依本研究所訂臨床試驗/研究計畫,因而發生不良反應造成損害,由長庚醫療財團法人林口長 庚紀念醫院與試驗主持人依法負補償責任。但本受試者同意書上所記載之可預期不良反應,不 予補償。
- (2)如依本研究所訂臨床試驗/研究計畫,因而發生不良反應或損害,長庚醫療財團法人林口長庚紀念醫院願意提供專業醫療照顧及醫療諮詢。您不必負擔治療不良反應或傷害之必要醫療費用。
- (3)除前二項補償及醫療照顧外,本研究不提供其他形式之補償;也未投保人體試驗責任保險。若您不願意接受這樣的風險,請勿參加試驗/研究。

頁 4 之 9

(4)您不會因為簽署本同意書,而喪失在法律上的任何權利。

十五、保護隱私與機密性

1.將會有一個研究代碼代表您的身分,此代碼不會顯示您的姓名、身分證字號、住址。

2.對於您訪查的結果及診斷,研究主持人將持保密的態度,小心維護您的隱私。如果發表研究養療財團

113. 4. 24



版本日期

果,您的身分仍將保密。

- 3.請您亦瞭解若簽署同意書即同意您的訪查紀錄可直接受監測者、稽核者、研究倫理委員會及主管機關檢閱,以確保本研究過程與數據符合相關法律及法規要求。上述人員並承諾絕不違反您的身分之機密性。
- 4.請您瞭解基於安全考量,研究團隊可能會告知或連繫您的其他科別主治醫師,使其了解您參與的 試驗及疾病治療狀況,以避免藥物交互作用造成危害。
- 5.由於試驗藥物同時在美國和歐盟進行試驗,依美國或歐盟藥品管理規定,則試驗結果將公佈於公開的臨床試驗資訊網站: Clinicaltrials.gov (美國), clinicaltrialsregister.eu (歐盟),但您的個人資料仍將保密,該網站只會有試驗之結果摘要,您可以在任何時候搜尋該網站。 (若不適用本段請刪除)

## 十六、試驗之退出與中止

受試者或立同意書人有權在無任何理由情況下,隨時要求終止參與試驗,此將不會減損您的正當醫療權益與法律權利。試驗主持人或贊助廠商亦可能於必要時中止該試驗之進行。

為了您的安全,當發生以下情形時,您必須退出試驗/研究:

- 1. 患者無法完成預定的 MRI 檢查
- 2. MRI 影像品質不足,無法定位臨床顯著攝護腺癌(csPCA)或排除 csPCA 的存在

當試驗/研究執行中有重要的新資訊(指和您的權益相關或是影響您繼續參與意願),會通知您並進一步說明,請您重新思考是否繼續參加,您可自由決定,不會引起任何不愉快或影響其日後醫師對您的醫療照顧。

當您退出本試驗或主持人判斷您不適合繼續參與本試驗時,在退出前已得到的資料將被保留,不會移除。

1.退出後讓試驗主持人繼續收集我的資料,例如經由我的病歷記載取得後續醫療過程、實驗室檢查結果。繼續收集資料期間,仍會維護您的隱私和個人資料的機密性。

□同意收集。

□不同意本試驗/研究繼續收集或檢視我的資料,但可經由公共資料庫查詢之紀錄不在此限。

## 十七、受試者權利

- 1.對於您個人資料之蒐集、處理及利用,試驗機構/試驗主持人將依受試者同意書、臨床試驗相關法 規及個人資料保護法相關規定辦理。您可以依據個人資料保護法之規定,以書面連絡試驗機構/試 驗主持人而行使下列權利:
  - (1)查詢或請求閱覽您的個人資料;
  - (2)請求提供您個人資料的影印本;
  - (3)請求補充或更正您的個人資料;
  - (4)請求停止蒐集、處理或利用您的個人資料;
  - (5)請求刪除您的個人資料。
- 2. 研究過程中,凡可能影響您繼續接受臨床試驗意願的任何重大發現,都將及時提供給您。研究過程中如有任何的問題或狀況,請與主持人聯繫。
- 3.對身為受試者之權利有意見或懷疑因參與研究而受害時,可與本院之人體試驗倫理委員會聯絡請求諮詢,其電話號碼為:(03)319-6200轉 3707、3703、3705~3709、3711~3714、3716~3717。

## 十八、試驗成果及權益歸屬

本研究預期不會衍生專利權或其他商業利益。

113 4 2

十九、個人資料、檢體與檢體衍生物之保存與再利用

長庚醫療財團法.



頁 5 之 9 版本日期

所有新的研究計畫都要再經由長庚醫療財團法人人體試驗倫理委員會審議通過,人體試驗倫理委員 會若認定新的研究超出您同意的範圍,將要求我們重新得到您的同意。 1. 個人資料 在試驗期間,依據試驗計畫類型與您所授權的內容,我們將會蒐集與您有關的病歷資料,並以一個 試驗編號來代替您的名字及相關個人資料。以電子方式儲存或建檔以供統計與分析之用,將會存放 於設有密碼與適當防毒軟體之專屬電腦內。文件資料將會統一保存於研究大樓6樓泌尿科實驗室。 數位資料將於保存至試驗正式停止後三年,屆時統一由計畫主持人馮思中醫師銷毀。 是否同意個人資料提供未來林口長庚紀念醫院研究之用,並授權長庚醫療財團法人人體試驗倫理委 員會審議是否需要再取得您的同意: □ 1.不同意保存我的個人資料,試驗結束後請銷毀 受試者簽名: 日期: 年 月 日 □ 2.同意以非去連結之方式保存我的病歷資料,逾越原同意使用範圍時,需再次得到我的同意才可 使用我的檢體進行新的研究,所有個人資訊及病歷資料將會保存至試驗正式停止後三年,屆 時將予以銷毀。 □我同意本次研究結束後的病歷資料,存入長庚醫療財團法人 長庚紀念醫院人體生物資料 庫,供後續其他經本院人體試驗倫理委員會核准之研究使用 (請同時簽署人體生物資料庫參 與者同意書)。 

## 二十、聲明

1.本試驗內容及同意書已經\_\_\_\_\_(請填寫取得同意書人姓名)完整口頭告知及說明,受試者本人/ 法定代理人已充分瞭解並同意,本同意書一式二份,已將研究用人體檢體採集同意書之副本交給受 試者。

> 人體試驗倫理委員會 核 准 日 期

113. 4. 24

長庚醫療財團法人

| A.受試者: | (正楷姓名) | | | | | |
|---|---|---|---|---|---|---|
| | (簽名) 日期: | 年月_ | 日 | | | |
| B.共/協同主持人: | (正楷姓 | (名) | | | | |
| | (簽名) | 日期:年_ | 月 | 日 | | |
| C.研究主持人: | (正楷姓名 | <b>7</b> ) | | | | |
| | (簽名)日 | 期:年 | _月日 | | | |
| **收案對象符合【同意書 | 簽署說明】第(一 | ·)項時,此欄位 | 必須簽名* | * | | |
| **主持人負有取得有效自 | 願性同意之義務 | ,需盡合理之努 | 力確認法 | 定代理人/有同意權人/監 | 護人 | |
| /輔助人之身分** | | | | | | |
| D.法定代理人/有同意權人 | /監護人/輔助人 | | | | | |
| **我已詳細閱讀以上資訊 | ,或者上述資訊 | 已由研究團隊人 | 員朗讀讓 | 我了解。我已有機會對之 | <b></b> 基研 | |
| 究提出問題,所提問題 | 亦已獲得詳細解 | 釋。我身為受試 | <b>活</b> 的 | | | |
| □配偶□父□母□兒□女 | □其他: | 我同意受試 | 【者參與本學 | 研究。** | | |
| (正楷姓. | 名) | | | | | |
| (簽名) □ | 日期:年 | _月日 | | | | |
| 電話: | | | | | | |
| **收案對象符合【同意書 | 簽署說明】第(二 | )項時,此欄位。 | 必須簽名** | <b>k</b> | | |
| E.見證人: | (正楷姓名) | | | | 人體試驗倫理委核 准 日 期 | A . |
| | (簽名)日期:_ | 年月 | 日 | | 113. 4. 24<br>長庚醫療財團 | |
| 長庚醫療財<br>CHANG GUNG MEDI | <b>国法人</b><br>CAL FOUNDATION | 頁7之9 | 版本日期 | 20240402 MRI v3 | | |

## 【同意書簽署說明】

## (一)法定代理人/有同意權人/監護人/輔助人使用時機:

- \*醫療法 第79條/人體研究法 第12條/藥品優良臨床試驗準則 第五條/研究用人體檢體採集注意事項 第6條:
- 1.受試者為無行為能力(未滿七歲之未成年人者或受監護宣告之人),由法定代理人為之;受監護宣告之人,由監護 人擔任其法定代理人。
- 2.受試者為限制行為能力者(滿七歲以上之未成年人或受輔助宣告之人),應得其本人及法定代理人或輔助人之同
- 会試者雖非無行為能力或限制行為能力者,但因意識混亂或有精神與智能障礙,而無法進行有效溝通和判斷時, 由有同意權之人為之。
- 4.採集胎兒之檢體,需經其母親同意。
- 5.屍體檢體之提供應得其最近親屬或本人生前之書面同意。

## (二)見證人使用時機:

- \*藥品優良臨床試驗準則 第二十一條:
- 1.受試者、法定代理人或有同意權人皆無法閱讀時,應由見證人在場參與所有有關受試者同意書之討論。見證人應 閱讀受試者同意書及提供受試者之任何其他書面資料,以見證研究主持人或其指定之人員已經確切地將其內容向 受試者、法定代理人或有同意權之人解釋,並確定其充分了解所有資料之內容。
- 2.受試者、法定代理人或有同意權人,仍應於受試者同意書親筆簽名並載明日期。但得以指印代替簽名。
- 3.見證人於完成口述說明,並確定受試者、法定代理人或有同意權人之同意完全出於其自由意願後,應於受試者同 意書簽名並載明日期。
- 4.研究相關人員不得為見證人。

### (三)法定代理人簽署順序:

\*依據醫療法第七十九條:醫療機構施行人體試驗時,應善盡醫療上必要之注意,並應先取得接受試驗者之書面同 意;接受試驗者以有意思能力之成年人為限。但顯有益於特定人口群或特殊疾病罹患者健康權益之試驗,不在此 限。

\*依據人體試驗管理辦法 第五條:依據醫療法第七十九條第一項但書召募之成年或已結婚未成年之受試者,主持人 應依下列順序取得其關係人至少一人之同意:

- 配偶。
- 二、 父母。
- 同居之成年子女。 三、
- 四、 與受試者同居之祖父母。
- 五、 與受試者同居之兄弟姊妹。
- 最近一年有同居事實之其他親屬。

前項第一款至第五款關係人之同意,以有同居事實者優先。

第一項關係人之同意,不得違反受試者曾表示之意思。

## 【長庚醫療財團法人長庚紀念醫院/長庚大學/長庚科技大學 研究參與者需知】

親愛的受試者、家屬、民眾,您好:

在您符合試驗或研究之納入條件時,您有可能會被邀請參與長庚醫院(長庚大學/長庚科技大學)的研究計畫,為了保 障您參與研究的安全與權益,以下內容將向您說明長庚醫療財團法人人體試驗倫理委員會所做的努力與把關,包含:研 究計畫如何審查、審查的重點為何以及受試者的權利。

#### ● 什麼是研究?

「研究」和「治療」是不一樣的。「治療」是已經歷經研究過程,完全了解治療以後可能發生的結果及副作用的發 生機率。但「研究」是為了解答我們原來所不知道的知識,並不完全清楚會發生怎樣的結果。因此,研究不是一定 要参加,且不参加不會影響您後續接受醫療照護的權益或者遭受任何不公平的待遇。

● 什麼是人體試驗倫理委員會?

「人體試驗委員會(Institutional Review Board,簡稱 IRB)」是為確保人體試驗或研究符合科學與倫理適當性,所設立 的審查單位。由具專業知識的醫療人員,及法律專家、社會公正人士或民間團體代表等非醫學背景人士組成,協助 研究人員了解受試者的處境,以確保受試者的安全與權益。**受試者對參與研究之相關權益有任何問題時,都可向長** 庚醫療財團法人人體試驗倫理委員會詢問。

▶ 人體試驗倫理委員會如何審查臨床試驗/研究計畫?審查的重點為何?

人體試驗倫理委員會 (1) 在長庚醫院(長庚大學/長庚科技大學)執行的研究,都需要經過長庚醫療財團法人人體試驗倫理委員會的審查,通 113. 4. 24 過了才可執行。

(2) 送到人體試驗倫理委員會的研究計畫,都會經過委員或者專家,以獨立、專業且謹慎的態度進行審查,審查的重以則表

長庚醫療財團法人 CHANG GUNG MEDICAL FOUNDATION

頁 8 之 9 版本日期

點,包含:是否有詳盡告知受試者試驗相關的事宜(包含:試驗目的、試驗進行程序等)、其他可能替代的治療方 式、參與研究的副作用、風險及好處、如何退出研究、參加者的照護與隱私是否受到保護等。

- (3) 在進行臨床研究審查時,長庚醫療財團法人人體試驗倫理委員會將評估這些研究計畫對於參與研究者可能造成的 風險有哪些?有些風險是屬於身體上的疼痛、不適,有些則帶來心理上的不舒服,有些甚至對於您的社會及經濟 方面造成影響,長庚醫療財團法人人體試驗倫理委員會就是要去確保這些風險帶來的傷害已經盡力降到最小。除 了風險,我們也會去評估參與研究者從研究中預期得到的好處、這項研究可能會治癒疾病、可能不會痊癒疾病但 可能改善受試者生活品質、或對參加的人可能不會有好處,但對醫學研究的進步或對未來患有相同疾病的人發現 新的治療方式而有所貢獻。長庚醫療財團法人人體試驗倫理委員會將**綜合評估每個研究計畫的風險相對於獲得的** 好處是不是合理,以決定是否通過該計畫,風險大而對受試者或科學知識沒有任何好處的研究,將不會通過人體 試驗倫理委員會的審查。
- (4) 研究計畫通過後,長庚醫療財團法人人體試驗倫理委員會與執行機構(長庚醫院/長庚大學/長庚科技大學),會針對 通過的計畫持續監督,以確定研究團隊確實按照通過的計畫書妥善執行,為受試者的權益把關。
- ▶ 做為一位受試者您的權利是什麼?
- ✓ 知的權利
  - (1)了解研究的目的是什麼?

研究人員應該以通俗易懂的話,告訴您這個研究的目的是什麼。

(2)研究過程將發生什麼事?

也就是您需要知道這個研究的程序該如何進行,包含:研究過程要您身上做哪些事?該怎麼配合?(例如隔多久 要回診一次?每次要抽多少血?做什麼檢查?),會帶給生活多少不便?

(3)不参加研究有沒有其他治療方法?

研究不是一定要參加,因此您有權知道是否還有其他治療方法。

(4)可能會發生什麼不良反應或風險?

任何研究一定有風險,因此需知道參加此研究的危險性有多大?同時,也務必了解萬一發生危險或緊急狀況時, 該怎麼辦?和誰聯絡?如何聯絡?以及誰會提供後續醫療救治?還有相關費用問題。在加入研究前,研究人員都 應仔細向您說明。

(5)參與研究可能帶來什麼好處與試驗預期的成果?

研究人員有義務向您說明,這個研究可能對您帶來的好處,或者這個研究可能不會直接對您受益,但研究成果可 能會發現新的治療方式對醫學進步、未來的人類有所貢獻,以便提供您考慮是否加入此研究。

(6)如果您想退出研究計畫,改如何提出?

研究人員應該告訴您,若您參加研究後中途想退出,應該向誰提出?退出後有無照護計畫?退出研究後,您在參 與期間所提供的資料是否繼續分析或保存?

- (7)當您有任何疑慮時,隨時可以向研究人員詢問
- 自由選擇參加研究的權利

在研究人員向您充分解釋研究目的、研究進行程序、其他可能的替代治療、參加研究可能遭遇的風險與帶來 的好處、研究的預期成果、退出試驗計畫的程序以及退出後的照護計畫後,經過您自主且有足夠時間的考慮是否 **参加此研究**,並且簽署受試者同意書,您才算正式加入研究,成為受試者。

此外,如果您想要退出研究,您可以於任何時間點,不需要任何的理由,向研究的相關人員提出。而您退出 的決定,也不會影響您後續接受醫療照護的權益或者遭受任何不公平的待遇。

#### ✓ 被保護的權利

(1) 隱私與機密的保護

對於您於參與研究期間所提供的任何資訊,研究團隊人員有義務維護您的隱私,如果發表研究成果,或為確保研 究過程與數據符合相關法律及法規要求,人體試驗倫理委員會或主管機關(例如:衛生福利部)將會檢閱研究之相 關資訊,但您的身分仍將被保密。

(2) 保有您現在所擁有的合法權利

參與臨床研究時,並不會放棄您的任何合法的權利。

人體試驗倫理委員會 核准日期

113. 4. 24

長庚醫療財團法人

長庚醫療財團法人 CHANG GUNG MEDICAL FOUNDATION

版本日期